CLINICAL TRIAL: NCT00516542
Title: A Phase I Study of DHEA in Combination With Letrozole in ER- Breast Cancer
Brief Title: Dehydroepiandrosterone (DHEA) and Letrozole in Treating Patients With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated due to lack of accrual
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOL-06019-L; R21CA119598 (NIH); P30CA069533 (NIH); OHSU-e2109; OHSU-IRB00002109
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Letrozole; Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: letrozole — A daily dose of 2.5 mg will be used throughout the study.
Drug: DHEA — Will be dispensed in either 500mg or 1000mg tablets. Subjects will start at a dose of 500 mg and may increase up to 5000mg depending on the cohort.
Other: pharmacological study — PK draws will happen on day 1 and day 14, then every 2 weeks.

SUMMARY:
RATIONALE: Androgens can cause the growth of breast cancer cells. Hormone therapy using dehydroepiandrosterone (DHEA) may fight breast cancer by blocking the use of androgen by the tumor cells. Letrozole may stop the adrenal glands from making androgens. Giving DHEA together with letrozole may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of DHEA when given together with letrozole in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the maximum tolerable dose, dose-limiting toxicity, and pharmacokinetics of dehydroepiandrosterone (DHEA) when given together with letrozole in patients with androgen receptor-positive and estrogen receptor- and progesterone receptor-negative metastatic breast cancer.

OUTLINE: Patients receive oral dehydroepiandrosterone and oral letrozole once daily. Physical exams and blood collections are performed every two weeks. Tumor assessments are performed once every three months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

  * Metastatic disease
* Hormone receptor status

  * Estrogen receptor- and progesterone receptor-negative
  * Androgen receptor-positive

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Postmenopausal (> 60 years of age)
* Leukocyte count > 3,000/uL
* Absolute neutrophil count > 1,500/uL
* Platelet count > 100,000/uL
* Total bilirubin normal
* AST and ALT < 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance > 60 mL/min

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior chemotherapy
* At least 4 weeks since prior biologic therapy
* At least 4 weeks since prior radiotherapy
* At least 30 days since prior investigational agents
* No concurrent dehydroepiandrosterone or androstenedione supplements
* No concurrent chemotherapy or radiotherapy
* No concurrent hormone therapy or immunotherapy (including trastuzumab [Herceptin®])

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | One year from drug start
  Subjects will be monitored at day 14 and then every 2 weeks for up to one year.

CONTACTS AND LOCATIONS:
Overall Officials: Rodney F. Pommier, MD, Study Chair — Oregon Health and Science University
Locations (1):
- Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon, United States